CLINICAL TRIAL: NCT00815321
Title: Autologous Cytokine Induced Killer Cells as Adjuvant Adoptive Immunotherapy in Patients With Chronic Myeloid Leukemia on Standard Drug Therapy
Brief Title: Autologous Cytokine Induced Killer Cells (CIK) for Chronic Myeloid Leukemia (CML) Patients on Standard Drug Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIK#3/2008
Record Dates: First submitted 2008-12-28; First posted 2008-12-30 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Chronic Myeloid Leukemia
Keywords: chronic myeloid leukemia; autologous cytokine induced killer cells; Chronic myeloid leukemia in blast crisis treated with chemotherapy or kinase inhibitors; Chronic myeloid leukemia with mutation resistant to kinase inhibitors; chronic myeloid leukemia with good response to kinase inhibitor and stable persistence of residual disease
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Autologous CIK cell infusion — 4 CIK cells will be infused into patients at regular 3-weekly intervals for 4 infusions. The target cell dose per infusion is 1x10e10 CD3 cells. For patients with uncontrolled accelerated or blastic transformation undergoing chemotherapy, this will be given at the nadir of lymphopenia following chemotherapy. For other patients this will be given without interruption of the ongoing treatment with Imatinib or other kinase inhibitor.

SUMMARY:
This is an extension of our ongoing clinical trial using ex vivo expanded autologous Cytokine-induced killer (CIK) cells as an adoptive cellular immunotherapy for haematological malignancies. The pre-existing clinical trial targets patient with acute myeloid leukemia or MDS, and relapsed disease post allogeneic transplant.

Chronic myeloid leukemia (CML) is a disease with good response to kinase inhibitors. There are however patients in transformed phase of the disease who do not respond to these treatment. A small proportion of patients with response to Imatinib may develop mutations resulting in drug resistance. In addition, the vast majority of patients with a good response to the kinase inhibitors still have persistent CML cells detectable at a molecular level. It is known that the CML progenitors are not sensitive to the kinase inhibitors. On the other hand, immune mediated mechanism is known to be able to eradicate CML as shown by efficacy of donor lymphocyte infusion in the allogeneic transplant setting. Early clinical trials have shown clearance of bcr-abl using peptide vaccination. There is also convincing mouse data showing eradication of CML at molecular level by autologous CIK cells, but no clinical trial has been done using CIK cells for CML.

We therefore plan to expand our current CIK trial to include CML as a disease, for CML patients with various degree of response to the kinase inhibitors which have already offered its maximal effect. We aim to study whether autologous CIK cells may further improve disease response, either in the eradiation of minimal residual disease, or in conjunction with chemotherapy for control of high tumour load disease.

DETAILED DESCRIPTION:
Patients with CML falls into various groups based on their disease stage and response to kinase inhibitors. In the context of currently available kinase inhibitors, allogeneic transplant and the various available new drug trials, there are still some patients who will not achieve a satisfactory or sustainable response. For such patients, we aim to employ CIK cell as an immunotherapeutic modality concurrent with their original CML-specific therapy. This will enable us to explore any additional activity of CIK cells against CML without any compromise to their ongoing, established treatment.

The following groups of patients are potential candidates:

1. Blast crisis / accelerated phase patients who have failed to response to the kinase inhibitors but are fit to undergo induction chemotherapy as for the acute leukemia. Repeated cycles of CIK will be given in phase with the planned chemotherapy cycles, to observe for achievement of any remission and its durability.
2. Blast crisis / accelerated phase patients who have achieved a haematological or cytogenetic response to the kinase inhibitors, but do not have further definitive curative options eg allogeneic transplant. In the absence of long term data with Dasatinib or Nilotinib , it is justifiable to study the efficacy of addition of CIK therapy to their baseline best response achievable with drug therapy.
3. Patients with resistance to the currently available kinase inhibitors due to T315I mutation or other undefined mutations, with progressive relapse either at molecular, cytogenetic or haematological level, and do not have transplant as a curative option. In this group of patients additional of CIK to current treatment will show any activity of CIK against the drug-resistant mutant CML cells.
4. Patients who have achieved a stable but residual molecular evidence of CML, who are willing to explore additional means with a hope to eradication of MRD. Since the role of immunotherapy is most relevant in MRD, CIK infusion will provide the proof of principal observation of whether imatinib-resistant CML Philadelphia stem cells can be eradicated by these ex vivo activated and expanded cytotoxic T cells.

ELIGIBILITY:
Inclusion Criteria:

1. Blast crisis / accelerated phase patients who have failed to response to the kinase inhibitors but are fit to undergo induction chemotherapy as for the acute leukemia.
2. Blast crisis / accelerated phase patients who have achieved a haematological or cytogenetic response to the kinase inhibitors, but do not have further definitive curative options
3. Patients with resistance to genetic or haematological level, and do not have transplant as a curative option.
4. Patients who have achieved a stable but residual molecular evidence of CML, who are willing to explore additional means with a hope to eradication of MRD.

Patients must understand the trial nature of this study and the additional leukapheresis procedure needed for harvesting mononuclear cells.

Exclusion Criteria:

On recruitment :

1. Renal impairment with Cr >200mmol/uL
2. Liver impairment with transaminase >5x upper limit which is not due to disease
3. Limited life expectancy <3 months

On day of infusion

1. uncontrolled infection or significant bleeding
2. unstable vital signs
3. any degree of hypoxia requiring oxygen therapy.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-12; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
response of CML to Cytokine induced killer cell therapy | 6 -12 months

SECONDARY OUTCOMES:
Sustainability of the response | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Yeh Ching Linn, MBBS, MRCP, Principal Investigator — Singapore General Hospital
Locations (1):
- Dept of Haematology, Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Background] Bhatia R, Holtz M, Niu N, Gray R, Snyder DS, Sawyers CL, Arber DA, Slovak ML, Forman SJ. Persistence of malignant hematopoietic progenitors in chronic myelogenous leukemia patients in complete cytogenetic remission following imatinib mesylate treatment. Blood. 2003 Jun 15;101(12):4701-7. doi: 10.1182/blood-2002-09-2780. Epub 2003 Feb 6. PMID 12576334
- [Background] Graham SM, Jorgensen HG, Allan E, Pearson C, Alcorn MJ, Richmond L, Holyoake TL. Primitive, quiescent, Philadelphia-positive stem cells from patients with chronic myeloid leukemia are insensitive to STI571 in vitro. Blood. 2002 Jan 1;99(1):319-25. doi: 10.1182/blood.v99.1.319. PMID 11756187
- [Background] Rousselot P, Huguet F, Rea D, Legros L, Cayuela JM, Maarek O, Blanchet O, Marit G, Gluckman E, Reiffers J, Gardembas M, Mahon FX. Imatinib mesylate discontinuation in patients with chronic myelogenous leukemia in complete molecular remission for more than 2 years. Blood. 2007 Jan 1;109(1):58-60. doi: 10.1182/blood-2006-03-011239. Epub 2006 Sep 14. PMID 16973963
- [Background] Kolb HJ, Schattenberg A, Goldman JM, Hertenstein B, Jacobsen N, Arcese W, Ljungman P, Ferrant A, Verdonck L, Niederwieser D, van Rhee F, Mittermueller J, de Witte T, Holler E, Ansari H; European Group for Blood and Marrow Transplantation Working Party Chronic Leukemia. Graft-versus-leukemia effect of donor lymphocyte transfusions in marrow grafted patients. Blood. 1995 Sep 1;86(5):2041-50. PMID 7655033
- [Background] Pinilla-Ibarz J, Cathcart K, Scheinberg DA. CML vaccines as a paradigm of the specific immunotherapy of cancer. Blood Rev. 2000 Jun;14(2):111-20. doi: 10.1054/blre.2000.0127. PMID 11012250
- [Background] Bocchia M, Gentili S, Abruzzese E, Fanelli A, Iuliano F, Tabilio A, Amabile M, Forconi F, Gozzetti A, Raspadori D, Amadori S, Lauria F. Effect of a p210 multipeptide vaccine associated with imatinib or interferon in patients with chronic myeloid leukaemia and persistent residual disease: a multicentre observational trial. Lancet. 2005 Feb 19-25;365(9460):657-62. doi: 10.1016/S0140-6736(05)17945-8. PMID 15721470
- [Background] Linn YC, Lau LC, Hui KM. Generation of cytokine-induced killer cells from leukaemic samples with in vitro cytotoxicity against autologous and allogeneic leukaemic blasts. Br J Haematol. 2002 Jan;116(1):78-86. doi: 10.1046/j.1365-2141.2002.03247.x. PMID 11841399
- [Background] Alvarnas JC, Linn YC, Hope EG, Negrin RS. Expansion of cytotoxic CD3+ CD56+ cells from peripheral blood progenitor cells of patients undergoing autologous hematopoietic cell transplantation. Biol Blood Marrow Transplant. 2001;7(4):216-22. doi: 10.1053/bbmt.2001.v7.pm11349808.
- [Background] Introna M, Borleri G, Conti E, Franceschetti M, Barbui AM, Broady R, Dander E, Gaipa G, D'Amico G, Biagi E, Parma M, Pogliani EM, Spinelli O, Baronciani D, Grassi A, Golay J, Barbui T, Biondi A, Rambaldi A. Repeated infusions of donor-derived cytokine-induced killer cells in patients relapsing after allogeneic stem cell transplantation: a phase I study. Haematologica. 2007 Jul;92(7):952-9. doi: 10.3324/haematol.11132. PMID 17606446
- [Background] Hoyle C, Bangs CD, Chang P, Kamel O, Mehta B, Negrin RS. Expansion of Philadelphia chromosome-negative CD3(+)CD56(+) cytotoxic cells from chronic myeloid leukemia patients: in vitro and in vivo efficacy in severe combined immunodeficiency disease mice. Blood. 1998 Nov 1;92(9):3318-27. PMID 9787169
- [Background] Li Z, Qiao Y, Liu B, Laska EJ, Chakravarthi P, Kulko JM, Bona RD, Fang M, Hegde U, Moyo V, Tannenbaum SH, Menoret A, Gaffney J, Glynn L, Runowicz CD, Srivastava PK. Combination of imatinib mesylate with autologous leukocyte-derived heat shock protein and chronic myelogenous leukemia. Clin Cancer Res. 2005 Jun 15;11(12):4460-8. doi: 10.1158/1078-0432.CCR-05-0250. PMID 15958631
- [Background] Leemhuis T, Wells S, Scheffold C, Edinger M, Negrin RS. A phase I trial of autologous cytokine-induced killer cells for the treatment of relapsed Hodgkin disease and non-Hodgkin lymphoma. Biol Blood Marrow Transplant. 2005 Mar;11(3):181-7. doi: 10.1016/j.bbmt.2004.11.019. PMID 15744236